CLINICAL TRIAL: NCT06910878
Title: Urinary Tract Infections Caused by Extended-spectrum Beta-lactamase-producing Enterobacteria: Management by General Practitioners in Bas-Rhin.
Brief Title: Urinary Tract Infections Caused by Extended-spectrum Beta-lactamase-producing Enterobacteria
Acronym: EBLSE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9307
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Urinary Tract Infections
Keywords: Urinary Tract Infections; Beta-Lactamase; Enterobacteriaceae
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary tract infections (UTIs) are one of the most common pathologies encountered in general practice. However, with increasing bacterial resistance to antibiotics, their treatment is becoming increasingly complex. Extended-spectrum beta-lactamase-producing Enterobacteriaceae (ESBL-E) pose a particular challenge due to their increased resistance to many commonly used antibiotics. The aim of this thesis is to study the management of such infections by general practitioners in Bas-Rhin and to suggest possible avenues for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Subject with an Enterobacteriaceae urinary tract infection treated in a primary care setting for urinary tract infection between June 1, 2024 and December 31, 2024
* Subject not objecting, after being informed, to the reuse of their data for the purposes of this research.
* The subject's primary care physician agreeing to participate in the study

Exclusion Criteria:

* Subject and/or their primary care physician having expressed their opposition to participating in the study
* Subject under legal protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years old) with an Enterobacteriaceae urinary tract infection treated in a primary care setting for urinary tract infection between June 1, 2024 and December 31, 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Prescription rates of appropriate antibiotics for the treatment of ESBL-E UTIs | Up to 1 year
  Prescription rates of appropriate antibiotics for the treatment of ESBL-E UTIs by general practitioners compared to current health authority recommendations

CONTACTS AND LOCATIONS:
Locations (1):
- Service de maladies infectieuses et tropicales - Hôpitaux Universitaires de Strasbourg, Strasbourg, France